CLINICAL TRIAL: NCT01505283
Title: Effect of Epidural Analgesia on the Parameter ANI During Childbirth
Acronym: APD-ANI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment difficulties
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2010/20; 2011-A00962-39 (Other: ANSM)
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain | interventions — Sodium Chloride; Sufentanil; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group Saline (Placebo Comparator): Epidural administration of saline
  Interventions: Drug: NaCl 0.9%
- Group Sufentanil (Experimental): Epidural administration of sufentanil
  Interventions: Drug: Sufentanil
- Group Lidocaine (Experimental): Epidural administration of lidocaine
  Interventions: Drug: lidocaine

INTERVENTIONS:
Drug: NaCl 0.9% — epidural administration of 6 ml of NaCl 0.9%
  Arms: Group Saline
Drug: Sufentanil — epidural administration of sufentanil 10 µg
  Arms: Group Sufentanil
Drug: lidocaine — epidural administration of lidocaine 50 mg
  Arms: Group Lidocaine

SUMMARY:
There are many methods used for the assessment of pain in the area of anesthesia including heart rate variability which reflects the influence of the autonomic nervous system on the heart. An original index, the ANI (Analgesia Nociception Index), quantifies pain during anesthesia. Obstetric epidural analgesia is particularly suited to evaluate ANI in conscious patients with a comparison of ANI with the measurement of pain by a visual analog scale (VAS).

Evaluation of ANI is performed just before epidural catheter insertion and during the 10 first minutes after saline, sufentanil or lidocaine epidural administration.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years,
* ASA I or II,
* No history of cardiovascular or respiratory disease
* No cardiovascular medication
* No treatment with a tocolytic agent(salbutamol, nicardipine)
* Desiring epidural analgesia at the early phase of labor pain

Exclusion Criteria:

* Too fast labour
* A pain score at or above 70 on the pain scale
* A disturbed EKG signal or extrasystoles
* Pace-Maker
* Diabetes mellitus

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2011-12; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Comparison of the ANI parameter with the VAS during labour | 2 hours
  The main objective of the research is to evaluate ANI as a measurment of pain caused by uterine contractions.

SECONDARY OUTCOMES:
Effects of epidural sufentanil and of epidural local anesthetic on ANI | 2 hours
  The secondary objective is to compare the effects of epidural sufentanil and a local anesthetic on the parameter ANI.
Effects of anxiety score on ANI | 2 hours
  The secondary objective is to study the effects of anxiety on the parameter ANI.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, MD, Study Chair — Hopital Foch; Morgan Le Guen, MD, Principal Investigator — Hopital Foch
Locations (1):
- Hopital Foch, Suresnes, Île-de-France Region, France